CLINICAL TRIAL: NCT06898476
Title: A Prospective, Double-Blind, Randomized Controlled Trial Evaluating Silkworm Pupa Powder Versus Placebo in Improving Alzheimer's Disease Among Patients
Brief Title: Silkworm Pupa Powder Improves Dementia.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Provincial Tongde Hospital (Other)
Collaborators: Hangzhou Institute of Medicine Chinese Academy of Sciences (Unknown)
Responsible Party: Principal Investigator, Jiangtao Zhang, Jiangtao Zhang, Chief Physician, Zhejiang Provincial Tongde Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Jiangtao Zhang
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease(AD); Sarcopenia; Asthenia
Keywords: Alzheimer Disease; Sarcopenia; asthenia; nutritional status; frailty state
MeSH Terms: conditions — Alzheimer Disease; Sarcopenia; Asthenia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Silkworm pupa powder, 2 times a day, two packets (12*2 g) each time, take with warm water, before meals, for three months
  Interventions: Dietary Supplement: Silkworm pupa powder
- Control group (Placebo Comparator): Placebo, 2 sachets (12*2 g) twice a day, with warm water, before meals, for three months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Silkworm pupa powder — Silkworm pupa powder, 2 times a day, two packets (12*2 g) each time, take with warm water, before meals, for three months
  Arms: Experimental Group
Dietary Supplement: Placebo — Placebo, 2 sachets (12*2 g) twice a day, with warm water, before meals, for three months
  Arms: Control group

SUMMARY:
The purpose of this clinical trial is to determine whether silkworm pupa powder is effective in treating Alzheimer's disease. It will also investigate whether silkworm pupa powder can improve the nutritional and frailty status of patients with Dementia. The main questions it aims to answer are:

* Will silkworm pupa powder improve the daily living conditions of patients with Alzheimer's disease?
* Will silkworm pupa powder improve the nutritional status and frailty of Alzheimer's disease patients?

Researchers will compare silkworm pupa powder with a placebo (a similar substance containing 0.5% silkworm pupa powder) to see if silkworm pupa powder can treat Alzheimer's disease.

Participants will:

* Take silkworm pupa powder or placebo daily for four months;
* Visit the clinic for check-ups and tests every four weeks;
* Record their symptoms and various physiological indicators.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's disease (AD) according to the National Institute on Aging-Alzheimer's Association (NIA-AA) criteria, with disease severity classified as mild, moderate, or severe (i.e., Mini-Mental State Examination [MMSE] total score between 0 and 24 points [inclusive] at screening and baseline).
* Confirmation of AD pathology per the 2024 revised AD diagnostic criteria (biomarker-defined AD with both Aβ and tau positivity):
* Aβ positivity: Plasma Aβ42/40 ratio ≤0.08 or amyloid-PET positivity (SUVR ≥1.1).
* Tau positivity: Plasma p-tau217 ≥2.5 pg/mL or CSF p-tau181/Aβ42 ratio ≥0.02.
* Age: 50 to 90 years of age (inclusive), with at least a primary school education. Both males and females are eligible.
* Stable medication use: If receiving approved AD therapies (e.g., acetylcholinesterase inhibitors, GV-971, NMDA receptor antagonists), doses must remain stable for ≥12 weeks prior to baseline. Treatment-naïve participants are also eligible. All other non-AD-related permitted concomitant medications must remain stable for ≥4 weeks prior to baseline unless otherwise specified.
* Hachinski Ischemia Scale (HIS) total score ≤4.
* Geriatric Depression Scale-15 (GDS-15) total score ≤4.
* Neuroimaging evidence: Screening CT/MRI showing age-related brain changes or cerebral atrophy.
* Caregiver availability: Participant has a stable and reliable caregiver, as confirmed by the investigator.
* Informed consent: Written informed consent must be provided by the participant or, if the participant lacks decision-making capacity, by a legally authorized representative (in accordance with local laws, regulations, and customs). Participants agree to provide peripheral blood, stool, and urine samples during the study for biomarker analysis.

Exclusion Criteria:

* Diagnosis of dementia other than Alzheimer's disease (AD) or other central nervous system disorders.
* Unstable vital signs accompanied by abnormalities in cardiac, pulmonary, hepatic, renal, or other organ functions.
* Abnormally low folate and/or vitamin B12 levels, or evidence that hypothyroidism has caused or exacerbated the participant's dementia. Participants with abnormal syphilis test results.
* Patients with comorbid psychiatric disorders.
* Long-term alcoholism or substance abuse that may compromise the evaluation of treatment efficacy.
* Participants with intolerance or allergy to the study medications.
* Abnormalities detected on cranial MRI, including ischemic or hemorrhagic infarctions, hydrocephalus, or brain tumors.
* Diagnosis of clinically significant cardiovascular or cerebrovascular disease requiring treatment within 12 months or at present.
* Antibiotic use:

  1. Continuous antibiotic use for more than 10 days within 12 weeks prior to baseline.
  2. Anticipated need for antibiotic treatment exceeding 10 days during the study.
* Geriatric Depression Scale-15 (GDS-15) score >4 at screening.
* Any other inadequately controlled condition (e.g., cardiac, respiratory, renal, or gastrointestinal disorders affecting absorption, such as gastric cancer, gastric bypass surgery, or recurrent diarrhea) that may jeopardize participant safety or interfere with study assessments, as judged by the investigator.
* Participation in any clinical trial involving novel chemical entities for Alzheimer's disease (AD) within 6 months prior to screening, unless confirmed to have been in the placebo group.
* Clinically significant abnormalities in physical examination, vital signs, laboratory tests, or electrocardiogram (ECG) requiring further investigation, treatment, or posing risks to study procedures/safety.
* Participation in clinical trials involving therapeutic monoclonal antibodies, antibody-derived proteins, immunoglobulin therapy, or vaccines within 6 months prior to screening, unless confirmed to have been in the placebo group.
* Participation in clinical trials involving anti-amyloid therapies (including monoclonal antibodies or BACE inhibitors), unless confirmed to have received only placebo.
* Uncontrolled immune disorders requiring treatment with immunoglobulins, systemic monoclonal antibodies (or derivatives), systemic immunosuppressants, or plasmapheresis during the study.
* Participants with uncontrolled bleeding disorders, including platelet count <50,000 or INR >1.5 (for those not on anticoagulants, e.g., warfarin). Participants on anticoagulants must have optimized and stable dosing for ≥4 weeks prior to screening. Anticoagulated participants are excluded from cerebrospinal fluid (CSF) assessments.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) | The 0th、 4th 、8th and 12th week after taking Silkworm
  The ADAS-Cog is a tool designed to assess the severity of cognitive impairment in patients with Alzheimer's disease (AD). It consists of 12 items that evaluate multiple cognitive domains, including memory, orientation, language, praxis (practical ability), attention, and others. Through a series of standardized cognitive tasks, it measures the severity of AD-related cognitive symptoms and tracks changes in response to treatment. Higher total scores indicate more severe cognitive impairment.
Frailty indicators | The 0th、 4th 、8th and 12th week after taking Silkworm Silkworm pupa powder.
  This study employs serum 25-hydroxyvitamin D concentration as the central biomarker for frailty assessment. The selection is predicated on vitamin D's pivotal role in preserving musculoskeletal function and neuroprotective mechanisms, coupled with established evidence that suboptimal 25-hydroxyvitamin D levels exhibit significant correlations with geriatric frailty syndrome and cognitive decline. Through quantitative analysis via high-precision mass spectrometry, dynamic monitoring of vitamin D status alterations pre- and post-intervention will be conducted. Further investigation will elucidate its associations with frailty phenotypes (e.g., grip strength, gait speed) and dementia progression pathways.
Frailty indicators | The 0th、 4th 、8th and 12th week after taking Silkworm Silkworm pupa powder.
  Plasma D-dimer concentration has been incorporated into the core biomarker panel for frailty assessment.Change in plasma D-dimer levels from baseline to 12 months, measured by immunoassay, to evaluate its association with disease progression in Alzheimer's disease

SECONDARY OUTCOMES:
Cognitive and Global Functional Assessment: | The 0th、 4th 、8th and 12th week after taking Silkworm Silkworm pupa powder.
  The combined evaluation of cognitive decline and global clinical status in Alzheimer's disease (AD) will be assessed using:
  Clinician's Interview-Based Impression of Change plus caregiver input (CIBIC-plus):
  A semi-structured clinician-rated scale capturing global changes in cognition, function, and behavior, incorporating caregiver perspectives.
  Mini-Mental State Examination (MMSE):
  A validated 30-point cognitive screening tool evaluating domains including orientation, memory, attention, language, and visuospatial abilities.
  Rationale:
  The dual assessment leverages:
  CIBIC-plus for holistic, clinician-judged disease progression (anchored to baseline severity).
  MMSE for quantifiable tracking of specific cognitive deficits. This approach aligns with FDA guidelines for multidimensional evaluation of therapeutic efficacy in AD trials (e.g., 21 CFR 314.510).
  Statistical Analysis:
  Changes in CIBIC-plus (ordinal scale) and MMSE scores (continuous scale) will be analyzed longitudinally,
Assessing patient nutritional improvement using Third Lumbar Skeletal Muscle Index (L3-SMI). | The 0th、 4th 、8th and 12th week after taking Silkworm Silkworm pupa powder.
  The nutritional index is evaluated using the Third Lumbar Skeletal Muscle Index (L3-SMI): A single cross-sectional image of L3 is obtained through CT scanning, and skeletal muscles in the image are identified and quantified using a HU threshold of -29 to 150. The total muscle area at this level is calculated using 3D Slicer software, and then divided by the square of the height (m^2) to obtain the Third Lumbar Skeletal Muscle Index (L3-SMI).
  Time Frame: The 0th、 4th 、8th and 12th week after taking Silkworm Silkworm pupa powder.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongde Hospital of Zhejiang Province, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided